CLINICAL TRIAL: NCT00509457
Title: Immunotherapy in Patients With Non-small Cell Lung Cancer (NSCLC). A Phase II Study of GV 1001 Telomerase Peptide Vaccination in Patients With Locally Advanced NSCLC
Brief Title: GV 1001 Immunotherapy in Patients With Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: St. Olavs Hospital (Other); Sorlandet Hospital HF (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-002646 11; 2006-50 DNR
Record Dates: First submitted 2007-07-20; First posted 2007-07-31 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2009-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: NSCLC, vaccination; Inoperable NSCLC stage IIIA/B in good performance status
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

INTERVENTIONS:
Biological: GV 1001 Telomerase peptide

SUMMARY:
To examine the safety and efficacy of telomerase peptide vaccination ( stimulation of the immune system) in patients with NSCLC after having been treated with conventional therapy with radiotherapy and docetaxel as a radiosensitizer.

DETAILED DESCRIPTION:
Survival in patients with locally advanced, inoperable NSCLC may be improved if local control can be achieved with concurrent chemo radiotherapy .After completed standard chemo-and radiation therapy; the safety and efficacy of vaccination therapy will be measured as time to progression after treatment with GV1001. Analysis of changes in T-cell subpopulations and cytokines in peripheral blood will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with inoperable NSCLC, disease stage IIIA and stage IIIB, who has received concurrent chemoradiotherapy( typically docetaxel 20 mg/m2 and 3D radiotherapy, 2Gy x 30 within the last 4 weeks.
* No sign of brain metastasis( excluded by MRI of the brain)
* Male or female above the age of 18 years.
* Normal lab. values

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-11; Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
To examine if combined chemoradiotherapy in patients with NSCLC followed by vaccination( immunotherapy) will increase the immunological response compared to previous experience

SECONDARY OUTCOMES:
Number of T cell responders and DTH responders, time to progression of disease

CONTACTS AND LOCATIONS:
Overall Officials: Steinar Aamdal, Principal Investigator — Oslo University Hospital
Locations (1):
- Rikshospitalet - Radiumhospitalet HF, Oslo, Norway